CLINICAL TRIAL: NCT06600945
Title: Atracurium Versus Atracurium and Magnesium Sulphate As Adjuvants to Local Anesthetic for Peribulbar Anesthesia in Cataract Surgery
Brief Title: Atracurium Versus Atracurium and Magnesium Sulphate As Adjuvants to Local Anesthetic
Status: Recruiting | Type: Observational
Sponsor: Dalia yousry Mohamed elsayed (Other)
Collaborators: Minia University (Other)
Responsible Party: Sponsor-Investigator, Dalia yousry Mohamed elsayed, Atracurium Versus Atracurium and Magnesium Sulphate as Adjuvants to Local Anesthetic for Peribulbar Anesthesia in Cataract Surgery, Minia University
Organization: Minia University (Other)
Other Study IDs: Peribulbar Anesthesia
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peribulbar Anesthesia
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Effect of addition of atracurium and magnesium sulphate to local anesthetic in peribulbar anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group c control group: Group C (Control group): Will undergo peribulbar block using 6ml of local anesthetic: 2ml of 0.5%bupivacaine and 1ml of 2% lidocaine mixed with hyaluronidase (150 U) + 2ml lidocaine 2 %+ 1ml 0.9% saline without atracurium and magnesium sulphate
  Interventions: Other: Cataract surgery
- Group A atracurium group: Group A (Atracurium group): Will undergo peribulbar block using 6ml of local anesthetic: 2ml of 0.5% bupivacaine and 1ml of 2% lidocaine mixed with hyaluronidase (150 U) + 2ml lidocaine 2%+ 0.05 mg/kg atracurium (maximum 5 mg) in 1 ml of 0.9% saline .
  Interventions: Other: Cataract surgery
- Group M magnesium sulphate group: Group M (Atracurium+ Magnesium sulfate): Will undergo peribulbar block using 6ml of local anesthetic: 2 ml of 0.5%bupivacaine and 1 ml of 2% lidocaine mixed with hyaluronidase (150 U) +2ml lidocaine2%+ (0.05 mg/kg atracurium (maximum 5 mg) + 50 mg magnesium sulfate) in 1 ml of 0.9% saline
  Interventions: Other: Cataract surgery

INTERVENTIONS:
Other: Cataract surgery — With local anesthetic in peribulbar anesthesia

SUMMARY:
To evaluate the effects of adding magnesium sulfate to atracurium with local anesthetic mixture on akinesia of globe and eyelid regarding onset and duration in cataract surgery using peribulbar technique

DETAILED DESCRIPTION:
Regional anesthesia is a preferred technique for ophthalmic surgery. It's safe, inexpensive and provides efficient ocular anesthesia for ophthalmic surgery.

Among regional blocks, peribulbar block is safe to retrobulbar block due to lesser incidence of series complications such as brain-stem anesthesia globe perfusion and retrobulbar hemorrhage .

The effect of non-depolarizing neuromuscular blockers on peribulbar anesthesia has been described in many studies. According to these studies the use of atracurium as adjuvant to peribulbar anesthesia provides early onset of akinesia and improves the quality of anesthesia in absence of any adverse effect.

Magnesium sulphate is non-competitive N-Methyl-D- Aspartate (NMDA) antagonism and calcium channel blocker. Magnesium has endothelium derived Nitric Oxide induced vasodilation. It enhanced the activity of local anesthetic agent and improves the quality of anesthesia .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cataract surgery (phacoemulsification and intraocular lens implantation).

Patients aged 20-80 years. Both sexes. ASA physical status I&II.

Exclusion Criteria:

- Refusal of the patient to participate in the study. Any disorder of neuromuscular system known from history or clinical examination e.g., Guillarian barre syndrome, Myasthenia gravies and Myopathies.

Patients are known to have a history of fits. Patients on medication known to interact with neuromuscular blocking drugs as antipyretics (aminoglycosides and tetracyclines), antiarrhythmic (quinidine).

Local sepsis. Coagulation abnormalities (INR>1.4). High myopia with axial length more than 30 mm or less than 21. Mentally retarded patients and failure of proper communication as in deafness. Morbidly obese patients (BMI>40). Patients with glaucoma (increased IOP>20mmgh). Patients with history of hypersensitivity to study drugs. Very dense or very soft cataract .

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both sexes and from 20 to 80 years
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Block quality | Baseline
  Occurance of motor and sensory block

SECONDARY OUTCOMES:
Block Success | Baseline
  Onset and duration of block.Post operative analgesia and pain score. Patient satisfaction and surgeon Satisfaction. Incidence of complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia yousry mohamed, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No